CLINICAL TRIAL: NCT00280774
Title: Memantine for Corticosteroid-Induced Mood and Declarative Memory Changes: A Pilot Study
Brief Title: Memantine for Corticosteroid-Induced Mood and Declarative Memory Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 102005-076; NAM-MD-26
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2007-07

CONDITIONS: Physiological Effects of Drugs
Keywords: corticosteroid; prednisone; memantine; Patients who are taking a corticosteroid for a; pulmonary illness; rheumatic illness; kidney transplant
MeSH Terms: interventions — Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
The purpose of this research is to determine if patients on corticosteroids who are given memantine will show improvement in memory compared to those receiving placebo (an inactive substance). This research also seeks to determine if such patients, when given memantine, will experience improvement in manic/hypomanic symptoms (feelings of agitation, overexcitement, or hyperactivity) and/or depressive symptoms. Subjects will be randomized to a crossover trial of memantine and placebo for 8 weeks, followed by a 4 week washout and then 8 more weeks of the study medication. Memantine and placebo will start at 5 mg/day for one week, increased to 5 mg twice a day in the second week. During the third week patients will take 10 mg in the morning and 5 mg in the evening. At weeks 4-8, patients will take 10 mg twice a day. One 8 week course of study medication will be memantine and the other 8 week course of study medication will be placebo, both assigned in a random fashion.

DETAILED DESCRIPTION:
Twenty (20) outpatients with pulmonary (e.g. asthma), rheumatic (e.g. rheumatoid arthritis, dermatomyositis) illnesses or renal transplants (all populations we have used in prior clinical trials) receiving a course of prednisone or other corticosteroid for at least 12 weeks will be enrolled. To participate, patients must be between the ages of 18 and 70 and taking at least 5 mg/day of prednisone, or a prednisone equivalent, for at least 3 months and with the expectation that they will be continuing such treatment at the same dose for at least 20 additional weeks. At baseline, the research assistant or study doctor will ask patients about their health, any prior corticosteroid therapy and other medications patients may take for any health problems, medication allergies, and any surgical procedures or cognitive impairments they may have. Patients will have memory tests and answer questions about their mood, sleep, appetite, and daily activities.

The subjects will be randomized to a crossover trial of memantine and placebo for 8 weeks followed by a 4 week washout and then 8 more weeks of study drug. Memantine will be started at 5 mg/day for 1 week, increased to 5 mg BID in the second week, 10 mg QAM and 5 mg QHS the next week and to 10 mg BID in weeks 4-8 as directed in the package insert. One 8 week course will be memantine and the other placebo assigned in a random fashion. Measures of memory will be compared within subjects at baseline, week 4, week 8, week 12 (beginning of second course of study drug), week 16 and week 20 (exit). At weeks 2 and 14, participants will be given 3 questionnaires that will measure mood; medication management will be conducted during these assessments. Each visit, including baseline, should take approximately one and a half hours.

Detailed Experimental: Baseline measures of mood will be assessed with the Activation subscale of the Internal State Scale (ISS) (primary measure), Hamilton Depression Rating Scale (17-item version), and Young Mania Rating Scale (YMRS). Cognition will be assessed with the HVLT-R (primary measure), and STROOP color word task. The subjects will be given memantine or identical appearing placebo as described above. Reductions in dosage will be allowed should clinically significant side effects emerge based on the judgment of a blinded psychiatrist. The above cognitive measures will be administered at each assessment visit (8 total); during the assessments at week 2 and week 14 patients will also be given 3 mood questionnaires. Each visit will be approximately an hour and half in length. The RA doing assessments will be blinded at all times. Alternative but equivalent versions of the HVLT-R will be given to minimize practice or learning effects. Current and cumulative corticosteroid dose (mg each day X number of days) will be determined and recorded.

In the case of missing data we will use the last observation carried forward. In our lamotrigine study in a similar population, we found a change in the total words recalled on a word list and on the Stroop. Assuming a similar change with memantine and using double-sided, paired t-tests, we could detect a difference with a change in the placebo group with participants on the HVLT-R and with participants on the STROOP. Thus, although this is primarily a pilot study to obtain effect sizes for future, larger trials funded by NIH, it should have power to detect clinically meaningful differences between medication and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients between (and including) ages 18-70 and taking at least 5 mg/day of prednisone equivalents for at least 3 months and anticipating continued treatment at the same dose for at least 20 additional weeks will be eligible for enrollment.

Exclusion Criteria:

* Patients with a history of allergic reaction or other contraindication to memantine therapy or with other unstable medical conditions (e.g. recent myocardial infarction, diabetes with poor glycemic control) will not be allowed to participate.
* Pregnant or nursing women or women of childbearing age who will not use University of Texas Southwestern (UTSW) Institutional Review Board (IRB) approved methods of avoiding pregnancy will be excluded from the study.
* Those with a history of mental retardation, dementia, or other severe cognitive disorders will also be excluded from the study.
* Patients with baseline RAVLT total words recalled normative score > 55 will be excluded to avoid including persons with exceptionally good declarative memory at baseline.
* Subjects who do not speak English will be excluded because many of the outcome measures used in this study are not validated in languages other than English.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
HVLT-R test total words recalled scores will be compared between baseline and exit of the active medication phase and placebo phase using a within subjects design and paired t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, Ph.D., M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System (Asthma, Allergy, & Arthritis Clinics), Dallas, Texas, United States

REFERENCES:
- [Derived] Brown ES, Vazquez M, Nakamura A. Randomized, placebo-controlled, crossover trial of memantine for cognitive changes with corticosteroid therapy. Biol Psychiatry. 2008 Oct 15;64(8):727-729. doi: 10.1016/j.biopsych.2008.05.010. Epub 2008 Jun 25. PMID 18582848